CLINICAL TRIAL: NCT06177236
Title: The Effect of in Clinic or Self- Sampling for Cervical Cancer Screening on Status of Particitipation, Attitude and Anxiety.
Brief Title: Clinic or Self-Sampling for Cervical Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, OZGE SEN, midwife, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: stanbulUC
Record Dates: First submitted 2023-11-22; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Cervical Cancer; HPV Infection
Keywords: cervical cancer; HPV testing
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- randomıze (Experimental): Assuming that a t-test between two independent groups with 80% power, d=0.5 effect size, and t-test between two independent groups will be used in the study, it was found that there should be at least 102 women in total, including 51 self-sampling and 51 clinician sampling groups. Considering the losses that may occur during the study, it was planned to include 110 women in the sample for this phase. These women will be randomly assigned to Self-Sampling (n=55) or Clinician Sampling (n=55) groups in a 1:1 ratio using https://randomizer.org/. The self-sampling group will be trained on the subject and will be provided with a self-sampling HPV DNA test kit, while the HPV DNA test
  Interventions: Diagnostic Test: cervical cancer screening

INTERVENTIONS:
Diagnostic Test: cervical cancer screening — The aim of this project was to determine the effect of clinic or self-sampling on attendance, attitudes, and anxiety in cervical cancer screening.

SUMMARY:
Objective: The aim of this project was to determine the effect of clinic or self-sampling on attendance, attitudes, and anxiety in cervical cancer screening.

DETAILED DESCRIPTION:
Introduction: Persistent infection with high-risk HPV strains is the main cause of cervical cancer.

Objective: The aim of this study was to determine the effect of clinic or self-sampling on cervical cancer screening participation, attitudes and anxiety in women.

Method: The study was conducted as a descriptive and randomized controlled study between October 2022 and December 2023 in Ödemiş ASM No. 2, Ministry of Health, Republic of Turkey. The first phase of the study was conducted with 309 women and the "Introductory Information Form" and "Attitude Scale for Early Diagnosis of Cervical Cancer" were used to evaluate participation and attitudes towards cervical cancer screening. The second phase of the study was conducted as a randomized controlled trial with 110 women in the experimental (n=55) and control (n=55) groups. The women in the experimental group were trained before the procedure and were allowed to take samples from the vaginal area on their own. The women in the control group were sampled from the cervical region by the clinician. Both groups were pretested before the procedure using the "Descriptive Information Form" and the "State Anxiety Inventory" to measure anxiety. After the sampling procedure, the post-test was administered to the experimental and control groups using the "State Anxiety Inventory".

Results: According to the screening method preferences of the women, 34% (n=105) preferred a self-test, 18.4% (n=57) preferred a test performed by a clinician in a clinic, 3.9% (n=12) preferred no method, and 43.7% (n=135) preferred both methods. In the study, it was found that the self-test option increased participation in screening. The mean total score of the women was found to be 102.896±5.660. This result shows that women have high positive attitudes towards early diagnosis of cervical cancer. In the second stage of the study, it was observed that the descriptive characteristics of the experimental and control groups showed homogeneous distribution. While there was no significant difference between the experimental and control groups in terms of anxiety level in the pretest, it was found that the control group had a significantly higher anxiety level in the posttest.

Conclusion: In this study, it was observed that women had positive attitudes towards cervical cancer screening, self-sampling increased participation in screening and decreased anxiety levels.

ELIGIBILITY:
Inclusion Criteria: Must be able to perform self-test

Exclusion Criteria: pregnancy, diagnosing the cervix

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 30-65 years old
Enrollment: 110 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
The Effect of in Clinic or Self-Sampling for Cervical Cancer Screening on Status of Participation | 1 year
  In the study, it was found that the self-test option increased participation in screening.

SECONDARY OUTCOMES:
The Effect of in Clinic or Self-Sampling for Cervical Cancer Screening on Status of ling for Cervical Cancer Screening on Status of Attitude | 1 year
  This result shows that women have high positive attitudes towards early diagnosis of cervical cancer.

OTHER OUTCOMES:
The Effect of in Clinic or Self-Sampling for Cervical Cancer Screening on Status of ling for Cervical Cancer Screening on Status of Anxiety | 1 year
  While there was no significant difference between the experimental and control groups in terms of anxiety level in the pretest, it was found that the control group had a significantly higher anxiety level in the posttest.

CONTACTS AND LOCATIONS:
Overall Officials: Özge Şen, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul Unıversıty-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No